CLINICAL TRIAL: NCT03320252
Title: Endurant CHevAr New Indication Trial: ENCHANT - Post-market Study of the Endurant CHEVAR Technique for the Treatment of Juxtarenal Aortic Aneurysms With a Short Infrarenal Neck
Brief Title: Endurant CHevAr New Indication Trial: ENCHANT
Acronym: ENCHANT
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT16022
Record Dates: First submitted 2017-09-21; First posted 2017-10-25 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: AAA - Abdominal Aortic Aneurysm
Keywords: CHEVAR; Chimney; Juxtarenal; Short Infrarenal /neck; Endurant
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endurant Chimney Graft Technique — Medtronic Endurant II and Endurant IIs Stent Graft Systems and balloon-expandable covered stent graft systems approved for use in the renal arteries. These devices will be utilized in a chimney graft configuration.

SUMMARY:
The purpose of the post-market study is to assess the clinical outcomes, safety, and performance of the Endurant Chimney Graft Technique (Endurant Stent Graft Systems used with a balloon-expandable covered stent graft) for treatment of juxtarenal aortic aneurysms with a short infrarenal neck in a real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years old
* Subject is scheduled for primary treatment of the juxtarenal aortic aneurysm with a short infrarenal neck (i.e. no revision subjects)
* Subject is able and willing to comply with the protocol and to adhere to the follow-up requirements
* Subject has provided written informed consent
* Subject is an eligible candidate according to the currently available Endurant II/IIs instructions for use for ChEVAR
* Subject has a juxtarenal aortic aneurysm with a short infrarenal neck (definition of juxtarenal aortic aneurysm with a short infrarenal neck will be in accordance with commercially available Endurant II/IIs instructions for use for ChEVAR).

Exclusion Criteria:

* Subject is participating in a concurrent study which may confound study results
* Subject has a life expectancy ≤ 2 year
* Subject has an aneurysm that is:

  * Suprarenal or pararenal
  * Isolated iliofemoral
  * Mycotic
  * Inflammatory
  * Pseudoaneurysm
* Subject requires emergent aneurysm treatment, for example, trauma or rupture
* Subject has previously undergone surgical treatment for abdominal aortic aneurysm
* Subject is a female of childbearing potential in whom pregnancy cannot be excluded
* Subject has a known hypersensitivity or contraindication to anticoagulants, anti-platelets, or contrast media, which is not amenable to pre-treatment
* Subject has a creatinine level >2.0 mg/dl (or >176.8 μmol/L) and/or is on dialysis
* Subject has an active COVID-19 infection or relevant history of COVID-19. Relevant history of COVID-19 is defined as availability of a positive COVID-19 test with sequela or hospitalization for treatment of COVID-19. Subjects with a positive COVID-19 test who were asymptomatic or had mild symptoms should be excluded only if the positive test was less than 6 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of subjects that meet the indications for the Endurant Chimney Graft Technique for the endovascular treatment of juxtarenal aortic aneurysms with a short infrarenal neck.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint evaluated by proportion of subjects experiencing a Major Adverse Event through 30 days post-index procedure | through 30 days post-index procedure
  Major Adverse Events include the occurrence of any of the following events:
  * All-cause mortality
  * Bowel ischemia
  * Myocardial infarction
  * Paraplegia
  * Procedural blood loss ≥1000 cc
  * Renal failure
  * Respiratory failure
  * Stroke
The primary performance endpoint is defined as the proportion of subjects who have technical success at the time of the index procedure and are free from secondary interventions through 365 days. | Index procedure and through 365 days

SECONDARY OUTCOMES:
Clinical Succes | Index procedure and within 30-days post-index procedure
  Technical success and freedom from intra-operative death and freedom from type Ia/III endoleak in the first image within 30-days post-index procedure
Secondary safety endpoints | through 30 days and annually up to 5 year follow up
  * Aneurysm rupture
  * Conversion to open surgery
  * Aneurysm related mortality
  * All-cause mortality
  * MAEs through 365 days
Secondary imaging based endpoints | at 30 days and at annual follow-up until 60 months post-index procedure
  * Stent graft fractures (endograft, chimney graft)
  * Stent graft occlusion (endograft, chimney graft)
  * Endoleak of all types
  * Stent graft migration >10 mm (endograft)
  * Aneurysm sac expansion ≥ 5 mm
Change in renal function | at 30 days and at annual follow-up until 60 months post-index procedure
  Change in renal function compared to baseline

CONTACTS AND LOCATIONS:
Locations (26):
- Ordensklinikum Linz GmbH / Elisabethinen, Linz, Austria
- France (2):
  - CHU de Bordeaux - Centre Universitaire Pellegrin, Bordeaux
  - Hôpitaux Universitaires Paris Ile-de-France Ouest - Hôpital Ambroise-Paré, Boulogne-Billancourt
- Germany (5):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Elisabeth Krankenhaus Essen GmbH, Essen
  - Universitäts Klinikum Frankfurt - Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Heidelberg, Heidelberg
  - St. Franziskus-Hospital Münster GmbH, Münster
- Greece (3):
  - Evaggelismos General Hospital of Athens, Athens
  - University Hospital of Larissa, Larissa
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
- Italy (3):
  - Azienda Ospedaliera di Cosenza, Cosenza
  - Ospedale Civile Sant'Andrea, La Spezia
  - Azienda Ospedaliera San Camillo Forlanini - Ospedale San Camillo, Roma
- Netherlands (3):
  - Stichting Rijnstate Ziekenhuis, Arnhem
  - Medisch Spectrum Twente, Enschede
  - Zuyderland Medisch Centrum, Heerlen
- Hospital de Santa Marta, Lisbon, Portugal
- Russian Cardiologic Research and Production Complex, Russian Ministry of Health, Moscow, Russia
- CINRE s.r.o., Bratislava, Slovakia
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Corporacío Parc Taulí - Hospital de Sabadell, Sabadell
- Skånes Universitetssjukhus Malmö, Malmo, Sweden
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
- United Kingdom (2):
  - St George's University Hospitals - NHS Trust, London
  - Central Manchester University Hospitals NHS - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No